CLINICAL TRIAL: NCT03622255
Title: Evaluation of Enamel Matrix Derivative as an Adjunct to Minimally Invasive Non-surgical Treatment of Intrabony Defects. A Randomized Controlled Clinical Trial.
Brief Title: Evaluation of Enamel Matrix Derivative as an Adjunct to Minimally Invasive Non-surgical Treatment of Intrabony Defects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Ioannis Vouros, Professor, Department of Preventive Dentistry, Periodontology and Implant Biology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09/23-11-2017
Record Dates: First submitted 2018-07-21; First posted 2018-08-09 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Periodontal Diseases
Keywords: Intrabony defects; Minimally invasive non-surgical technique; Enamel Matrix Derivative
MeSH Terms: conditions — Periodontal Diseases | interventions — emerin

STUDY DESIGN:
Intervention Model Description: A software (www.randomizer.org) will be used by one of the investigators who will not participate in the clinical and radiographic measurements nor the therapeutic intervention, to generate a block randomization. Thus, participants will be randomized in one of the two groups in a way that there is no difference between the two groups regarding the initial depth of the intrabony defect. In patients with more than one intrabony defects meeting the inclusion criteria, a second randomization scheme with the same software will take place, to determine which will be included. The randomization results will be placed in sealed envelopes accessible only to the principal investigator and opened for each patient after the end of MINST to determine if EMD will be applied or not.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINST (Other): Minimally invasive non-surgical technique (MINST): Root instrumentation under local anesthesia using specific hand instruments (micro- curettes) and delicate piezon ultrasonic instruments in the area of intraosseous defect.
  Interventions: Procedure: MINST
- MINST with EMD (Active Comparator): Minimally invasive non-surgical technique (MINST) with application of Enamel Matrix Derivative (EMD): Root instrumentation under local anesthesia using micro- curettes and delicate piezon ultrasonic instruments in the area of intraosseous defect. Experimental intervention by application of EDTA gel for 2 minutes on the root surface of the involved tooth, followed by rinsing with saline, drying and application of Enamel Matrix Derivative gel, to fill the defect.
  Interventions: Procedure: MINST with EMD

INTERVENTIONS:
Procedure: MINST — Minimally invasive non-surgical technique (MINST) for the treatment of intrabony defects has been compared with minimally invasive surgical treatment of these defects and has shown to achieve similar beneficial clinical results. In this study MINST will be used as the control treatment.
  Arms: MINST
Procedure: MINST with EMD — Enamel matrix derivative (EMD) has been widely used in the surgical treatment of periodontal intrabony defects, using a minimally invasive surgical technique (MINST). Recent studies have suggested that this product could also be used in the non-surgical treatment of intrabony defects using a minimally invasive technique with very good results. This study will evaluate the effect of enamel matrix derivative in the non-surgical treatment of periodontal intrabony defects when a minimally invasive technique is used. Besides clinical measurements, radiographic analysis will also be performed to evaluate the treatment results.
  Arms: MINST with EMD

SUMMARY:
Aim:

The aim of this prospective, randomized, parallel arm, blind, controlled clinical trial is to compare the clinical and radiographic outcomes following regenerative treatment of intrabony periodontal defects using a Minimally Invasive Non-Surgical Technique (MINST) with or without the application of Enamel Matrix Derivative (EMD)

Research Hypothesis:

The hypothesis is that the adjunctive application of EMD will enhance the clinical and radiographic results of minimally invasive non- surgical treatment of intrabony defects. Radiographic bone fill will be the primary outcome of the research, whereas CAL gain and PD reduction will constitute the secondary outcomes.

DETAILED DESCRIPTION:
Introduction Intrabony defects occur frequently in periodontitis and represent sites that, if left untreated, are at increased risk for disease progression. Although resective or repair procedures have been used to treat intrabony defects, aiming at their elimination, the treatment of choice is surgical periodontal regeneration. Over the last 30 years, histological and clinical studies have greatly improved our knowledge regarding regeneration of the periodontium and much attention has been given in clinical practice on the utilization of the principle of guided tissue regeneration (GTR), bone replacement grafts, biologics or their combination. Biologic factors appear attractive to alleviate local ⁄systemic factors counteracting periodontal wound healing ⁄ regeneration and untoward effects of biomaterials and devices as they become key components of novel regenerative technologies. The material most extensively researched as of today is enamel matrix derivative (EMD), which was first introduced in 1997.

Development of periodontal regeneration in the last 30 years has followed two distinctive, though totally different paths. The interest of researchers has so far focused on regenerative materials and products, on one side, and, on novel surgical approaches on the other side. In the area of materials and products, three different regenerative concepts have been mainly explored namely, barrier membranes, bone grafts, and wound healing modifiers, plus many combinations of the aforementioned. In the area of the surgical approaches, clinical innovation in flap design and handling as well as minimally invasive approaches has radically changed regenerative surgery.

In 1995, Harrel et al. introduced the first technical proposal of minimally invasive periodontal regenerative surgery (MIS) of isolated intrabony defects, with the aim to reduce surgical trauma, increase post-operative clot stability, improve flap adaptation and decrease time of surgery. Utilization of micro- surgical instruments and magnification was also proposed to minimize the trauma of the surgical procedure. The combination of this minimally invasive technique with EMD was also suggested by the same authors with successful long- term results.

Cortelini and Tonetti in 2007 presented a modification of the MIS technique. The authors proposed access of the defect- associated interdental papilla either with the modified papilla preservation technique- MPPT or the simplified papilla preservation technique- SPPT, depending on the width of the interdental space in combination with the application of EMD (MIST). Two years later, the same authors suggested a more tissue conservative technique, the modified- MIST (M-MIST). The surgical approach of M- MIST consists of a tiny intrasulcular incision performed only on the buccal side of the defect- associated tooth, which is connected with a horizontal incision performed as close as possible to the papilla tip. The palatal/lingual papilla are left untouched. In addition, Trombelli et al. suggested the single flap approach (SFA) in which a small incision is also performed only either buccally or palatially/lingually of the defect. Several randomized clinical trials published thereafter, comparing the efficacy of these minimally invasive techniques with or without the addition of regenerative factors, revealed equal results for both approaches, raising a series of hypotheses that focus more on the intrinsic healing potential of a wound when ideal conditions are provided with the surgical approach rather than the additive effect of regenerated material. Regenerative factors may increase the clot's initial stability and lead to better clinical results without though statistical significance.

More recently, a minimally invasive non- surgical technique (MINST) for treatment of intrabony defects was proposed. Initial clinical trials indicated comparable results to the surgical minimally invasive techniques in both clinical and microbiological outcomes. Considerable clinical and radiographic improvements after the application of MINST were also reported in a retrospective study, supporting its efficacy for treatment of intrabony defects. Additionally, an investigation designed to compare the effectiveness of EMD in combination with the MINST or MIST procedure in periodontal regeneration of deep intrabony defects concluded that the flapless procedure may be successfully applied in deep intrabony defects reaching clinical outcomes comparable with those of minimally invasive surgical approaches. So far, investigations comparing the outcomes of MINST as monotherapy or in combination with the use of EMD are missing. Thus, the purpose of this research is to compare the effectiveness of MINST with or without application of EMD in the treatment of intrabony defects.

Aim:

The aim of this prospective, randomized, parallel arm, blind, controlled clinical trial is to compare the clinical and radiographic outcomes following regenerative treatment of intrabony periodontal defects using a Minimally Invasive Non-Surgical Technique (MINST) with or without the application of Enamel Matrix Derivative (EMD)

Research Hypothesis:

The hypothesis is that the adjunctive application of EMD will enhance the clinical and radiographic results of minimally invasive non- surgical treatment of intrabony defects. Radiographic bone fill will be the primary outcome of the research, whereas CAL gain and PD reduction will constitute the secondary outcomes.

Procedure Before initiation of the study, the protocol will be approved by the Ethics Committee of the Dental School of the Aristotle University of Thessaloniki. In addition, informed consent will be signed by all participants.

Prior to inclusion in the study, an initial examination will be performed, including medical history, full- mouth plaque and bleeding scores, and PDs and CALs at 6 points on each tooth. In addition, oral hygiene instructions and motivation will be given. Patients will receive a supragingival debridement with ultrasonic instruments, in one session, without local anesthesia. Two weeks later a re-evaluation visit will be performed, including full- mouth plaque and bleeding scores and re-motivation to maintain proper oral hygiene. Four weeks after the initial visit (2 weeks after the first reassessment), the re- evaluation visit will be repeated. If the patient maintains appropriate oral hygiene levels (FMPS, FMBS <20%) he/she will be included in the study. If the bleeding and plaque scores are > 20%, a third re-evaluation visit will take place 2 weeks later (6 weeks after the initial visit) and if the scores reach the desired level, the patient will be included in the study. A software (www.randomizer.org) will be used by one of the investigators who will not participate in the clinical and radiographic measurements nor the therapeutic intervention, to generate a block randomization. Thus, participants will be randomized in one of the two groups in a way that there is no difference between the two groups regarding the initial depth of the intrabony defect. In patients with more than one intrabony defects meeting the inclusion criteria, a second randomization scheme with the same software will take place, to determine which will be included. The randomization results will be placed in sealed envelopes accessible only to the principal investigator and opened for each patient after the end of MINST to determine if EMD will be applied or not.

* Group A: application of minimally invasive non-surgical technique (MINST) for the intrabony defect and conventional non- surgical periodontal treatment in the rest of the quadrant teeth.
* Group B: application of minimally invasive non- surgical technique (MINST) with additional use of Enamel Matrix Derivative (EMD) for the intrabony defect and conventional non- surgical periodontal treatment in the rest of the quadrant teeth.

Treatment Procedures Group A: Minimally invasive non-surgical treatment (MINST). Root instrumentation under local anesthesia using specific hand instruments (micro- curettes) and piezon ultrasonic instruments in the area of intraosseous defect and scaling and root planing using conventional ultrasonic tips and hand instruments in the rest of the quadrant teeth.

Group B: Minimally invasive non-surgical treatment with application of enamel matrix derivative. Root instrumentation under local anesthesia using micro- curettes and piezon ultrasonic instruments in the area of intraosseous defect. Application of EDTA gel for 2 minutes on the root surface of the involved tooth. Rinsing with saline, drying and application of EMD to fill the defect. Scaling and root planing with conventional ultrasonic tips and hand instruments in the rest of the quadrant teeth.

Treatment in the remaining quadrants will proceed as following: the quadrant of the intrabony defect as well as the quadrant that will be in the same side of the mouth (either left or right) will be treated the same day with the MINST therapy. Both quadrants of the contralateral side will be treated in another day within the same week.

Treatment procedures will be performed with the use of 3.0 magnification and fiber optic lighting in both groups.

At the end of the treatment procedure, patients will be given instructions for use of a soft toothbrush without the additional use of interdental cleaning and use of 0.12% chlorhexidine solution (2 times a day) for 2 weeks. Two weeks after therapy, interdental cleaning will start with the adjunctive use of chlorhexidine gel 0.2% once a day for the first two weeks and 3 times a week for the rest of the study. Re-evaluation at 2 and 4 weeks, and 2, 3, 6, and 12 months will be scheduled. During these appointments FMPS and FMBS will be evaluated, oral hygiene instructions will be given and supragingival debridement will be performed when indicated. Clinical and radiographic measurements will be recorded at the 6th and 12th month examination.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age with a diagnosis of periodontitis.
* Have at least one isolated interproximal intrabony defect on a single-rooted tooth or a mandibular molar not extending to the furcation area with radiographic depth ranging between 3 mm-7 mm, pocket depth and clinical attachment loss ≥6 mm and radiographic defect angle ≤ 35o
* Proper oral hygiene: full-mouth plaque score (FMPS) ≤20% και full-mouth bleeding score (FMBS) ≤20%
* Systemically healthy (absence of systemic conditions that can affect the treatment outcome of periodontal therapy)

Exclusion Criteria:

* Pregnant or lactating female
* Current acute infection
* Non- surgical periodontal treatment the last 6 months or surgical periodontal treatment the last 12 months
* Teeth having an improper endodontic therapy with clinical signs of infection or subgingival restorations
* Tooth mobility 2nd- 3rd degree
* History of radiation therapy in the head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Radiographic bone fill | Change from baseline to 12 months
  Bone level in the intrabony defect

SECONDARY OUTCOMES:
Clinical attachment gain | Change from baseline to 12 months
  Clinical attachment level of intrabony defect measured in millimeters
Pocket depth reduction | Change from baseline to 12 months
  Pocket depth of intrabony defect measured in millimeters

OTHER OUTCOMES:
Recession | Change from baseline to 12 months
  Recession depth calculated as the difference of clinical attachment level minus probing depth.
Full mouth plaque score | Change from baseline to 12 months
  Percentage of tooth sites with detectable plaque
Full mouth bleeding score | Change from baseline to 12 months
  Percentage of tooth sites with bleeding when a periodontal probe is traced along the gingival margin
Distance from the CEJ or the margin of a restoration to the bottom of the defect (CEJ-BD) | Change from baseline to 12 months
  Measured in millimeters
Distance from the Cementoenamel Junction to the bone crest (CEJ-BC) | Change from baseline to 12 months
  Measured in millimeters
Depth of the intraosseous defect | Change from baseline to 12 months
  Distance from the bone crest to the bottom of the defect (BC-BD) measured in millimeters
Angle of the intraosseous defect | Change from baseline to 12 months
  Angle will be determined by the line defined by the root surface of the involved tooth and the line defined by the bone wall of the defect

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Vouros, DDS, Ph.D, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, School of Dentistry, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papapanou PN, Wennstrom JL. The angular bony defect as indicator of further alveolar bone loss. J Clin Periodontol. 1991 May;18(5):317-22. doi: 10.1111/j.1600-051x.1991.tb00435.x. PMID 2066446
- [Background] Susin C, Wikesjo UM. Regenerative periodontal therapy: 30 years of lessons learned and unlearned. Periodontol 2000. 2013 Jun;62(1):232-42. doi: 10.1111/prd.12003. PMID 23574469
- [Background] Darby IB, Morris KH. A systematic review of the use of growth factors in human periodontal regeneration. J Periodontol. 2013 Apr;84(4):465-76. doi: 10.1902/jop.2012.120145. Epub 2012 May 21. PMID 22612370
- [Background] Cortellini P. Minimally invasive surgical techniques in periodontal regeneration. J Evid Based Dent Pract. 2012 Sep;12(3 Suppl):89-100. doi: 10.1016/S1532-3382(12)70021-0. PMID 23040341
- [Background] Miron RJ, Sculean A, Cochran DL, Froum S, Zucchelli G, Nemcovsky C, Donos N, Lyngstadaas SP, Deschner J, Dard M, Stavropoulos A, Zhang Y, Trombelli L, Kasaj A, Shirakata Y, Cortellini P, Tonetti M, Rasperini G, Jepsen S, Bosshardt DD. Twenty years of enamel matrix derivative: the past, the present and the future. J Clin Periodontol. 2016 Aug;43(8):668-83. doi: 10.1111/jcpe.12546. Epub 2016 May 28. PMID 26987551
- [Background] Heijl L, Heden G, Svardstrom G, Ostgren A. Enamel matrix derivative (EMDOGAIN) in the treatment of intrabony periodontal defects. J Clin Periodontol. 1997 Sep;24(9 Pt 2):705-14. doi: 10.1111/j.1600-051x.1997.tb00253.x. PMID 9310876
- [Background] Hammarstrom L. Enamel matrix, cementum development and regeneration. J Clin Periodontol. 1997 Sep;24(9 Pt 2):658-68. doi: 10.1111/j.1600-051x.1997.tb00247.x. PMID 9310870
- [Background] Harrel SK, Rees TD. Granulation tissue removal in routine and minimally invasive procedures. Compend Contin Educ Dent. 1995 Sep;16(9):960, 962, 964 passim. PMID 8598026
- [Background] Harrel SK, Wilson TG, Nunn ME. Prospective assessment of the use of enamel matrix proteins with minimally invasive surgery. J Periodontol. 2005 Mar;76(3):380-4. doi: 10.1902/jop.2005.76.3.380. PMID 15857071
- [Background] Harrel SK, Wilson TG Jr, Nunn ME. Prospective assessment of the use of enamel matrix derivative with minimally invasive surgery: 6-year results. J Periodontol. 2010 Mar;81(3):435-41. doi: 10.1902/jop.2009.090393. PMID 20192871
- [Background] Cortellini P, Tonetti MS. A minimally invasive surgical technique with an enamel matrix derivative in the regenerative treatment of intra-bony defects: a novel approach to limit morbidity. J Clin Periodontol. 2007 Jan;34(1):87-93. doi: 10.1111/j.1600-051X.2006.01020.x. PMID 17243998
- [Background] Cortellini P, Prato GP, Tonetti MS. The modified papilla preservation technique. A new surgical approach for interproximal regenerative procedures. J Periodontol. 1995 Apr;66(4):261-6. doi: 10.1902/jop.1995.66.4.261. PMID 7782979
- [Background] Cortellini P, Prato GP, Tonetti MS. The simplified papilla preservation flap. A novel surgical approach for the management of soft tissues in regenerative procedures. Int J Periodontics Restorative Dent. 1999 Dec;19(6):589-99. PMID 10815597
- [Background] Cortellini P, Tonetti MS. Improved wound stability with a modified minimally invasive surgical technique in the regenerative treatment of isolated interdental intrabony defects. J Clin Periodontol. 2009 Feb;36(2):157-63. doi: 10.1111/j.1600-051X.2008.01352.x. PMID 19207892
- [Background] Trombelli L, Simonelli A, Pramstraller M, Wikesjo UM, Farina R. Single flap approach with and without guided tissue regeneration and a hydroxyapatite biomaterial in the management of intraosseous periodontal defects. J Periodontol. 2010 Sep;81(9):1256-63. doi: 10.1902/jop.2010.100113. PMID 20528696
- [Background] Cortellini P, Tonetti MS. Clinical and radiographic outcomes of the modified minimally invasive surgical technique with and without regenerative materials: a randomized-controlled trial in intra-bony defects. J Clin Periodontol. 2011 Apr;38(4):365-73. doi: 10.1111/j.1600-051X.2011.01705.x. Epub 2011 Feb 8. PMID 21303402
- [Background] Ribeiro FV, Casarin RC, Palma MA, Junior FH, Sallum EA, Casati MZ. Clinical and patient-centered outcomes after minimally invasive non-surgical or surgical approaches for the treatment of intrabony defects: a randomized clinical trial. J Periodontol. 2011 Sep;82(9):1256-66. doi: 10.1902/jop.2011.100680. Epub 2011 Feb 2. PMID 21284549
- [Background] Ribeiro FV, Casarin RC, Palma MA, Junior FH, Sallum EA, Casati MZ. Clinical and microbiological changes after minimally invasive therapeutic approaches in intrabony defects: a 12-month follow-up. Clin Oral Investig. 2013 Sep;17(7):1635-44. doi: 10.1007/s00784-012-0855-5. Epub 2012 Oct 5. PMID 23053707
- [Background] Nibali L, Pometti D, Chen TT, Tu YK. Minimally invasive non-surgical approach for the treatment of periodontal intrabony defects: a retrospective analysis. J Clin Periodontol. 2015 Sep;42(9):853-859. doi: 10.1111/jcpe.12443. Epub 2015 Sep 29. PMID 26257238
- [Background] Aimetti M, Ferrarotti F, Mariani GM, Romano F. A novel flapless approach versus minimally invasive surgery in periodontal regeneration with enamel matrix derivative proteins: a 24-month randomized controlled clinical trial. Clin Oral Investig. 2017 Jan;21(1):327-337. doi: 10.1007/s00784-016-1795-2. Epub 2016 Apr 5. PMID 27044318
- [Derived] Anoixiadou S, Parashis A, Vouros I. Enamel matrix derivative as an adjunct to minimally invasive non-surgical treatment of intrabony defects: A randomized clinical trial. J Clin Periodontol. 2022 Feb;49(2):134-143. doi: 10.1111/jcpe.13567. Epub 2021 Nov 9. PMID 34708441